CLINICAL TRIAL: NCT02181647
Title: Safe Touches: A Rigorous Evaluation of a Sexual Abuse Prevention Program for Children
Acronym: Safe Touches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The New York Society for the Prevention of Cruelty to Children (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R21HD069628 (NIH)
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Child Sexual Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Safe Touches Personal Safety Training for Children
  Interventions: Behavioral: Safe Touches: Personal Safety Training for Children
- Comparison (Other): Received Safe Touches after week-1 assessment completed (delayed intervention).
  Interventions: Behavioral: Safe Touches: Personal Safety Training for Children

INTERVENTIONS:
Behavioral: Safe Touches: Personal Safety Training for Children — The intervention includes a 50-minute interactive training and an age-appropriate activity book on personal body safety to take home and complete with caregivers. Using culturally appropriate puppets, workshop facilitators use role-play to model scenarios to help children: a) recognize safe and not-safe touches, b) understand body safety, c) practice assertiveness skills, and d) help children identify whom they can go to for help.

SUMMARY:
The primary goal of the study is to conduct a rigorous evaluation of the sexual abuse prevention program entitled, "Safe Touches: Personal Safety Training for Children (Safe Touches)." The main study hypothesis is that children who receive the Safe Touches intervention will show greater improvement on their knowledge of inappropriate touches compared to children who do not receive the intervention.

DETAILED DESCRIPTION:
This study will conduct a rigorous evaluation of the sexual abuse prevention program entitled, "Safe Touches: Personal Safety Training for Children (Safe Touches)." Founded in 2007, Safe Touches was developed for kindergarteners through third graders, and is conducted in the New York City public school system. The main goal of Safe Touches is to empower children to have personal agency over their bodies thus decreasing the likelihood of being inappropriately sexually touched and increasing the likelihood of disclosure if sexual abuse occurs.

While prior research provides some data regarding the efficacy of school-based child sexual abuse (CSA) prevention programs, evidence is profoundly marginal. First, most studies were not designed for multicultural populations, and therefore cannot inform what is effective in populations as diverse as New York City. A review of 22 studies evaluating school-based CSA prevention programs found just eight studies that used ethnically diverse samples, only one of which used a randomly assigned concurrent control group--however, this study had a very small sample size. Further, only three of the studies explored the mediating effects of factors such as gender and ethnicity on outcomes. The authors of those studies recommend future research that includes diverse samples and investigates differences in child characteristics more systematically--these recommendations are incorporated into the design and analysis plan of the current study. Second, statistical methods applied to data from prior studies were limited. A meta-analysis of 15 randomized controlled trials (RCTs) of school-based CSA prevention programs found that 10 studies used statistical analyses inappropriate for their particular design, thus increasing the risk for bias. Further, none of the 15 RCTs reported using the intention-to-treat principle. Third, no prior research has evaluated the cost of these programs relative to what children learn. In light of how common these programs are and the lack of valid evidence as to their efficacy, this study will determine their relative value with regard to acquisition of protective skills by addressing the first and second methodological gaps mentioned above, and expanding the scope to include the third, cost-effectiveness.

Study aims are:

1. To determine the significance of the difference in effectiveness between the Intervention and Control groups with regard to changes in children's recognition of unsafe touches/situations/people and acquisition of self-protective skills (short-term retention).
2. To evaluate maintenance of knowledge gains four weeks after intervention (maintenance).
3. To assess intervention costs relative to short-term retention and maintenance four weeks after intervention.

ELIGIBILITY:
Inclusion Criteria:

* second and third graders at participating New York City public schools
* at least 7 years old
* have not participated in Safe Touches program in the past

Exclusion Criteria:

* physical, cognitive, or emotional impairment that would affect the child's ability or safety in participating in the workshop or to respond to the questionnaire.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2012-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Children's Knowledge of Abuse Questionnaire | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary L. Pulido, Ph.D., Principal Investigator — The New York Society for the Prevention of Cruelty to Children
Locations (1):
- New York Society for the Prevention of Cruelty to Children, New York, New York, United States